CLINICAL TRIAL: NCT00647465
Title: Randomized Double-Blind Placebo Controlled Study Evaluating the Effect of Sublingual Administration of IFNa on the Immune Response to Influenza Vaccination in Subjects Aged 75 or More.
Brief Title: Effect of the Interferon Alpha Citizen by Sub-Lingual Way on the Humoral Immunizing Answer
Acronym: GP-INFA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: End of the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Orakine Ltd, Dublin, Ireland (Unknown)
Responsible Party: Mathieu QUINTIN, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P050601
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2005-11

CONDITIONS: Influenza Infection
Keywords: Influenza vaccine; interferon; adjuvant; the elderly
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): IFNalpha 2b
  Interventions: Drug: vaccine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vaccine — IFNalpha 2b
  Other Names: Influenza vaccination
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Influenza vaccination reduces the morbidity and mortality associated with influenza infection in at risk groups including the elderly and individuals with an impaired immune response, but is not totally protective in all recipient. Cytokines including type I interferons are known to play a key role in the innate immune response to virus infection and in the induction of the primary adaptive-immune response. Thus, we evaluated the safety of sublingual administration of IFNa and its effect on immune response to influenza vaccination in a randomized double-blind placebo controlled study in elderly institutionalized individuals.

DETAILED DESCRIPTION:
The protection afforded by the commonly used influenza sub-unit vaccines is thought to be due principally to the production of antibodies to viral haemagglutinin. The haemagglutination inhibitory (HAI) antibody titer is generally used as a surrogate marker of protection and a HAI antibody titer of 1:40 or greater is considered to confer protection. This is attained, however, in only 50% of elderly subject. Thus, there is an unmet need for an effective non-toxic adjuvant capable of enhancing the antibody response to influenza and other vaccines. Type I IFNs have been shown to induce B-lymphocytes to differentiate into antibody producing plasma cells and to be necessary for the production of both specific and polyclonal IgGs in response to influenza infection. Furthermore, type I IFNs increase the primary antibody response to a soluble antigen in vivo, and increase the production of all IgG sub-classes. Type I IFNs play a key role in adjuvant-induced Th1 responses. Thus, we evaluated the safety of sublingual administration of IFNa and its effect on immune response to influenza vaccination.Institutionalized subjects, aged 75 or more, were randomly assigned to two groups to receive in a double-blind fashion either 107 IU of Intron ATM in 1 ml of isotonic saline or 1 ml of saline alone (placebo) administered sublingually. Interferon or placebo were retained in the mouth for at least 30 seconds prior to ejection. All subjects were then vaccinated, within 30 minutes, with a single intramuscular injection (im) of influenza vaccine (InfluvacTM, Solvay Pharma, France).

The primary objective of this study is to compare the immunogenicity percentage of subjects who increased up to 4 fold their HAI antibody titer at day 21) obtained in the IFN treated group relative to the placebo treated group.

The secondary objectives are to compare mean HAI antibodies titers obtained in the two groups at day 21 ; specific IgG, IgG2a, IgG2a/IgG1 ratio and secretory IgA titers in the 2 groups; specific secretory IgA titers in saliva; durability of protective HAI antibodies titers 3 and 6 months after the vaccination and the safety of sublingual administration of IFNa.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 75 or more, -institutionalized-
* Subjects who were informed of the objectives of the study and who have given their written consent.
* Subjects who have received at least one prior influenza vaccination in the previous 5 years.
* Subjects who should be vaccinated against influenza during the 2005 vaccination campaign.

Exclusion Criteria:

* Individuals with severe disease, including neoplasia, autoimmune disease, or type I diabetes
* concomitant treatment with glucocorticoid or immunosuppressive drugs splenectomy or tonsillectomy
* or incapacity to open the mouth

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects presenting an increase > 4 fold of antiH1N1 or antiH3N2 or anti-B haemagglutination inhibition antibody titer, 3 weeks following influenza vaccination. | 21 days

SECONDARY OUTCOMES:
geometric mean of haemagglutination antibody titer obtained at day 21 with or without IFNa | 21 days
influenza virus strain-specific IgG total, IgG2a, IgG2a/IgG1 ratio, secretory IgA responses at day 21 in each group . | 21 days
influenza virus strain-specific secretory IgA anti-influenza antibody titers in saliva 14 and 21 days following vaccination. | 21 days
evaluation of individual response to IFNa treatment | 21 days
levels of serologic alpha interferon and of anti- alpha -interferon at day 21. | 21 days
Percentage of patients maintaining protective antibody titers 3 and 6 months following vaccination. | 3 months and 6 months after
Predictive factors of vaccine response (age, total lymphocyte cell count, CD4 cell count…) | 21 days
Evaluation of cellular vaccine response in a subgroup of subjects. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Bloch, MD, PhD, Principal Investigator — Assistance Publique-Hôpitaux de Paris, Groupe Hospitalier Broca-La Rochefoucauld, Service de Gérontologie 1 AP-HP
Locations (1):
- Assistance Publique-Hôpitaux de Paris, Groupe Hospitalier Broca-La Rochefoucauld, Service de Gérontologie 1, Paris, France